CLINICAL TRIAL: NCT02079662
Title: Integrative Oncology Program in Improving Cancer-Related Outcomes in Patients With Stage II or III Breast Cancer Undergoing Radiation Therapy
Brief Title: The Role of Lifestyle Factors in Breast Cancer-Related Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-0112; NCI-2014-02449 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0112 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (IO interventions) (Experimental): Patients undergo up to 7 different IO intervention sessions per week during their 6-week course of radiotherapy for between 1 and 3 hours each session, in addition to, up to 6 aerobic training sessions per week and one grocery store trip during the course of the program. IO intervention programs consist of nutritional coaching, behavioral therapy, yoga and meditation practice, resistance training, and a weekly meal sharing and cooking class. Patients then have weekly meetings with the study psychologist on the computer for 6 months, followed by a monthly meeting on the computer from 6-12 months, and 2 hour meetings at all follow-up appointments during the first year after radiotherapy.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Cognitive Intervention; Other: Computer-Assisted Intervention; Other: Counseling; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (standard of care) (Active Comparator): Patients undergo standard of care.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Behavioral, Psychological or Informational Intervention — Undergo IO intervention
  Arms: Arm I (IO interventions)
Other: Best Practice — Undergo standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard of care)
Other: Cognitive Intervention — Undergo IO intervention
  Arms: Arm I (IO interventions)
Other: Computer-Assisted Intervention — Undergo IO intervention
  Arms: Arm I (IO interventions)
Other: Counseling — Undergo counseling
  Other Names: Counseling Intervention
  Arms: Arm I (IO interventions)
Behavioral: Exercise Intervention — Undergo IO intervention
  Arms: Arm I (IO interventions)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies an integrative oncology (making changes in lifestyle and behavior) program in improving cancer-related outcomes in patients with stage II or III breast cancer undergoing radiation therapy. An integrative oncology program consisting of dietary recommendations, physical activity, stress management, social support, and control of environmental contaminants may modify cancer-related biological processes, influence long-term treatment results, and improve the quality of life of patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether the Integrative Oncology group (IO) has increased disease-free survival (time to recurrence) than the standard of care control group (SC).

II. Compare group differences over time in biological pathways including: immune function, endocrine function, insulin and glucose metabolism, cancer-related pathways (from peripheral blood), antioxidant capacity, and nutrient levels.

III. Examine group differences in overall survival. IV. Compare group differences over time in dietary patterns and fitness levels. V. Determine whether the IO group has improved patient reported outcomes including fatigue, sleep disturbances, radiotherapy toxicity (dermatitis, skin ulceration, pruritis, etc.), gut microbiome, other aspects of Quality of Life (QOL), mental health, social support, and measures of positive growth.

VI. Compare group differences over time in heart rate variability. VII. Determine cost-effectiveness analysis and work and/or home productivity.

SECONDARY OBJECTIVES:

I. Compare group differences over time in healthy breast tissue biomarkers acquired from fine needle aspirations.

II. Compare group differences in spouse or caregiver work productivity.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo up to 7 different IO intervention sessions per week during their 6-week course of radiotherapy for between 1 and 3 hours each session, in addition to, up to 6 aerobic training sessions per week and one grocery store trip during the course of the program. IO intervention programs consist of nutritional coaching, behavioral therapy, yoga and meditation practice, resistance training, and a weekly meal sharing and cooking class. Patients then have weekly meetings with the study psychologist on the computer for 6 months, followed by a monthly meeting on the computer from 6-12 months, and 2 hour meetings at all follow-up appointments during the first year after radiotherapy.

ARM II: Patients undergo standard of care.

After completion of study treatment, patients are followed up at 6 and 12 months and then annually for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage II or III breast cancer that will be scheduled to undergo a 4 to 6-week course of radiotherapy
* Participants must be able to read, write, and speak English
* Participants must be oriented to person, place, and time
* Participants must also meet at least two of the following criteria related to lifestyle: 1) consume less than 3 servings of fruit and vegetable/day; 2) engage in less than 75 minutes moderate/vigorous activity per week, defined as anything that causes small increases in breathing or heart rate for a sustained amount of time (e.g., brisk walking, bicycling); and 3) engage in a mind-body practice less than 4 times a month
* Participants must have a body mass index (BMI) of 24.45 or higher as assessed in the medical record

Exclusion Criteria:

* Patients with a recurrent breast cancer diagnosis
* Patients with another primary cancer diagnosis within 5 years of consent, not including non-melanoma skin cancers
* Patients who have any major psychiatric diagnoses or thought disorder (e.g. schizophrenia, bi-polar disorder, dementia)
* Patients with communication barriers (e.g., hard of hearing)
* Patients with extreme mobility issues (e.g. unable to get in and out of a chair unassisted)
* Patients with poorly or uncontrolled diabetes in the opinion of the physician(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Up to 5 years
  Will analyze DFS, using a multivariate comparison of DFS for each group using a Cox proportional hazards analysis. Will consider the following as potential covariates in the analysis (tumor and nodal status, menopausal status at diagnosis, tumor factors, treatment regimen, etc). Will obtain estimates for hazards ratios and 95% confidence intervals for the effect of the study arm and each covariate.
Changes in biological pathways | Baseline to 5 years
  Will use generalized linear mixed model regression (GLMM). Separate sets of analyses will be conducted for each criterion variable. To select the best method for modeling the repeated measures, will use the methods of Wolfinger and statistics such as Akaike's and Schwarz's information criteria. Will also use either t tests or Wilcoxon two-sample tests to analyze these data, depending on their distributions.
Changes in dietary patterns | Baseline to 5 years
  Will use GLMM. Separate sets of analyses will be conducted for each criterion variable. To select the best method for modeling the repeated measures, will use the methods of Wolfinger and statistics such as Akaike's and Schwarz's information criteria. Will also use either t tests or Wilcoxon two-sample tests to analyze these data, depending on their distributions.
Changes in fitness levels | Baseline to 5 years
  Will use GLMM. Separate sets of analyses will be conducted for each criterion variable. To select the best method for modeling the repeated measures, will use the methods of Wolfinger and statistics such as Akaike's and Schwarz's information criteria. Will also use either t tests or Wilcoxon two-sample tests to analyze these data, depending on their distributions.
Changes in heart rate variability | Baseline to 5 years
  Will use GLMM. Separate sets of analyses will be conducted for each criterion variable. To select the best method for modeling the repeated measures, will use the methods of Wolfinger and statistics such as Akaike's and Schwarz's information criteria. Will also use either t tests or Wilcoxon two-sample tests to analyze these data, depending on their distributions.
Changes in quality of life (including fatigue and sleep disturbances) | Baseline to 5 years
  Will use GLMM. Separate sets of analyses will be conducted for each criterion variable. To select the best method for modeling the repeated measures, will use the methods of Wolfinger and statistics such as Akaike's and Schwarz's information criteria. Will also use either t tests or Wilcoxon two-sample tests to analyze these data, depending on their distributions.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org